CLINICAL TRIAL: NCT02542644
Title: Assessment of Corneal Graft Attachment in Patients With Fuchs Endothelial Corneal Dystrophy Following Descemet's Membrane Endothelial Keratoplasty Using Ultra-high Resolution Optical Coherence Tomography
Brief Title: Assessment of Corneal Graft Attachment in Patients With Fuchs Endothelial Corneal Dystrophy Following DMEK Using Ultra-high Resolution OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-013015
Record Dates: First submitted 2015-08-31; First posted 2015-09-07 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Fuchs' Endothelial Dystrophy
Keywords: Fuchs' Endothelial Dystrophy, DMEK
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Fuchs endothelial dystrophy scheduled for DMEK (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT

INTERVENTIONS:
Device: Ultrahigh resolution Spectral Domain OCT — The area of graft detachment will be measured by a customized ultra high-resolution OCT for the cornea.
  A spectrometer based ultrahigh resolution Spectral Domain OCT (SDOCT) system operating at 800 nm for the anterior chamber will be employed in the present study. The spectrum of the Ti:Sapphire laser light source is centered at 800 nm. With a full width at half maximum bandwidth of 170 nm, the axial resolution is 1.3 μm in the cornea. The transverse resolution of the employed OCT system is 21 μm at the front surface of the cornea. For measurement, patients will place their head in a modified slit lamp head rest. During the measurement period, patients will be asked to look straight forward onto an internal fixation target and to avoid blinking. Different scattering patterns, e.g. raster, circular and spiral scans will be employed.

SUMMARY:
Fuchs endothelial corneal dystrophy (FECD) is a progressive disease characterized by the loss of endothelial cells, thickening of Descemet's membrane and deposition of extracellular matrix in the form of guttae. This result in failure of the endothelium to support corneal deturgescence leading to corneal edema. Affected patients complain about blurred vision at early stages of the disease which can progress to blindness. The pathophysiology of the disease is still unclear, but several studies point towards a genetic susceptibility. Additional risk factors that have been identified are female sex, smoking and older age.

While for a long time penetrating keratoplasty (PKP) was the only therapy available for affected patients, in the recent years less invasive methods such as descemet's membrane endothelial keratoplasty (DMEK) have been developed. In DMEK, only the Descemet's membrane and the endothelium is removed and replaced with the corresponding parts from a donor's cornea. For FECD, this brings the advantage that only the diseased part of the cornea is replaced. Graft detachment has been identified as the main complication following DMEK.

In the investigators' study, an ultra high resolution OCT system will be used to detect graft detachment in patients with FECD after DMEK. With this technique, even small detachments can be visualized. The area of graft detachment will be evaluated at predefined time points after surgery and correlated to visual acuity. A follow-up of one year will be performed in order to investigate the predictive value of graft adherence status at several time points for visual outcome.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years scheduled for primary DMEK because of Fuchs' Endothelial Dystrophy

Exclusion Criteria:

* Any disease inhibiting OCT acquisition; such as blepharospasm, severe tremor or immobility
* Any previous intraocular surgery other than cataract extraction
* Previous clinically significant ocular trauma in the study eye, as judged by the investigator
* Pregnancy, planed pregnancy, or lactating
* Appointment of a custodian
* Progressive retinal disease
* History or presence of glaucoma

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in best corrected visual acuity at 12 months compared to baseline using a standardized protocol with the Early Treatment Diabetic Retinopathy (ETDRS) charts (4 meters). | 1-2 days, 1 week, 1 month, 6 months and 12 months after DMEK
  Visual acuity will be measured using a standardized protocol with the Early Treatment Diabetic Retinopathy (ETDRS) charts (4 meters).
Area of attached graft after DMEK | 12 months after DMEK

SECONDARY OUTCOMES:
Number of patients in which rebubbling has to be performed | 12 months
Number of patients needing retreatment | 12 months
Best corrected visual acuity at 6 months using a standardized protocol with the Early Treatment Diabetic Retinopathy (ETDRS) charts (4 meters). | 6 months
  Visual acuity will be measured using a standardized protocol with the Early Treatment Diabetic Retinopathy (ETDRS) charts (4 meters).
Central corneal thickness | 12 months
Corneal endothelial cell count | 12 months
Demographic risk factors such as age | 12 months
Demographic risk factors such as gender | 12 months
Demographic risk factors, such as family history | 12 months
Demographic risk factors, such as smoking status | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Witkowska, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University Vienna, Department of Clinical Pharmacology, Vienna
  - Vienna Institute for Research in Ocular Surgery (VIROS), Vienna